CLINICAL TRIAL: NCT02818335
Title: Relative Bioavailability and the Effect of Food on the Bioavailability of LY3023414 in Healthy Subjects
Brief Title: A Study of LY3023414 Formulations and the Effect of Food
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 15696; I6A-EW-CBBB (Other: Eli Lilly and Company)
Record Dates: First submitted 2016-06-28; First posted 2016-06-29 (Estimated); Last update posted 2016-11-04 (Estimated); Status verified 2016-11

CONDITIONS: Healthy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- LY3023414 Reference Fasted (Experimental): Single oral dose of LY3023414 (Reference) on day one fasting.
  Interventions: Drug: LY3023414 Reference Fasted
- LY3023414 Test Fasted (Experimental): Single oral dose of LY3023414 (Test) on day one fasting.
  Interventions: Drug: LY3023414 Test Fasted
- LY3023414 Test Fed (Experimental): Single oral dose of LY3023414 (Test) on day one after a meal.
  Interventions: Drug: LY3023414 Test Fed

INTERVENTIONS:
Drug: LY3023414 Reference Fasted — Administered Orally
  Arms: LY3023414 Reference Fasted
Drug: LY3023414 Test Fasted — Administered Orally
  Arms: LY3023414 Test Fasted
Drug: LY3023414 Test Fed — Administered Orally
  Arms: LY3023414 Test Fed

SUMMARY:
The purpose of this study is to measure how much LY3023414 (a test formulation and a reference formulation) gets into the blood stream and how long it takes the body to get rid of it.

The study will also evaluate the effects of a high fat meal on LY3023414 compared to taking LY3023414 on an empty stomach. In addition, the tolerability of the study drug formulations will be evaluated. Information about any side effects that may occur will be collected.

This study includes 3 periods. Participants will be admitted to the clinical research unit (CRU) one day before dosing in each period. Total study duration is about 21 days, including follow-up. Screening may occur up to 30 days before the first dose of study drug.

This study is for research purposes only and is not intended to treat any medical conditions.

ELIGIBILITY:
Inclusion Criteria:

* Healthy surgically sterile or postmenopausal females and sterile males
* Have a body mass index (BMI) between 18.5 and 32.0 kilograms per meter squared (kg/m²), inclusive at screening

Exclusion Criteria:

* Cannot be investigative site personnel directly affiliated with this study or their immediate families. Immediate family is defined as a spouse, biological or legal guardian, child, or sibling
* Cannot be Lilly employees
* Have known allergies to LY3023414, related compounds, or any components of the formulation
* Regularly use known drugs of abuse and/or show positive findings on urinary drug screening
* Show evidence of human immunodeficiency virus (HIV) infection and/or positive human HIV antibodies
* Show evidence of hepatitis C and/or positive hepatitis C antibody
* Show evidence of hepatitis B and/or positive hepatitis B surface antigen

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07; Primary Completion 2016-10 (Actual); Study Completion 2016-10 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetics (PK): Area under the concentration versus time curve (AUC) from time zero to infinity (AUC[0-inf]) of LY3023414 | Pre-dose through 2 days post-dose in each period
Pharmacokinetics (PK): Area under the concentration from time zero to time t, where t is the last time point with a measurable concentration (AUC [0-tlast]) of LY3023414 | Pre-dose through 2 days post-dose in each period
Pharmacokinetics (PK): Maximum observed drug concentration (Cmax) of LY3023414 | Pre-dose through 2 days post-dose in each period
Pharmacokinetics (PK): Observed time of maximum concentration (tmax) | Pre-dose through 2 days post-dose in each period

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (1):
- Covance Clinical Research Inc, Daytona Beach, Florida, United States